CLINICAL TRIAL: NCT03360877
Title: Assessing the Risk of Hospital-acquired Infection and Multi-drug Resistance Among Hospitalized Severe Acutely Malnourished Children
Brief Title: Prevention of Nosocomial Infections (CleanKids)
Acronym: CleanKids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Minisitry of Public Health, Niger (Unknown); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NE-949
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Severe Acute Malnutrition; Health Care Associated Infection; Multi Drug Resistant Organisms
MeSH Terms: conditions — Severe Acute Malnutrition; Cross Infection

STUDY DESIGN:
Intervention Model Description: The initial 8-month baseline period will be used to collect data on the evaluation criteria of interest prior to the administration of any intervention of the study and will develop appropriate pedagogical tools to support the uptake of each cleaning strategy during subsequent intervention periods. After the reference period, a one-month introductory period will allow the organization of the first intervention at each site (ie - a soap and water cleansing administered by the carers in a structure or - a cleaning HCG administered by caregivers in the other facility) followed by eight months of active follow-up of the study with the first intervention. Following the eight months of active follow-up with the first intervention, there will be a crossover with an introductory period of one month and eight months of active follow-up with the other intervention. A final period of interruption will occur during the last eight months of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health-care associated infection (Other)
  Interventions: Other: Health-care associated infection (HCAI)

INTERVENTIONS:
Other: Health-care associated infection (HCAI) — Cleaning of the child with soap and water administered by the child's accompanying person in a structure or - a cleaning of the child with chlorhexidine gluconate administered by the child's accompanying person in the other structure

SUMMARY:
While the standardization of treatment protocols for Severe Acute Malnutrition (SAM) has helped to reduce historically high mortality, mortality in inpatient settings remains substantial, likely due to the severity of complications associated with late presentation and health-care associated infection (HCAI).

The purpose of this study is to serve as an important stand-alone description to inform the understanding of the magnitude of the problem and help guide implementation of measures to reduce the risk of nosocomial infection and multi-drug resistance.

DETAILED DESCRIPTION:
This study is designed as a cross-sectional, non-randomized, two-site, four-phase study: an initial baseline period, two intervention periods, and a final interruption period.

This is a descriptive study to collect information on the risk of HCAIs in the MSF-supported inpatient nutritional treatment centers. Information on key clinical indicators will be collected regularly according to the routine program procedures from the time of admission to discharge. All children will undergo a blood draw for culture at time of admission and at the time of any suspected hospital-acquired bloodstream infection. As part of active surveillance for bacterial colonization, including multi-drug resistant organisms, all children will undergo nasal and rectal swabs at the time of admission, suspected infection, and discharge. Data will provide an estimate of nosocomial infection incidence under routine circumstances and inform sample size calculations if further study is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. 6 to 59 months old
2. severe acute malnutrition with medical complications
3. parent / caregiver signing written informed consent

Exclusion Criteria:

1. health condition that does not allow blood draw
2. contraindication to the use of soap or Chlorhexidine gluconate, as recommended by the product
3. refusal to discontinue the use of skin care products that are incompatible with Chlorhexidine gluconate according to the product's directions for use

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4944 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the reduction of the incidence of nosocomial bacteremia | Between 48 hours after hospitalization and less than 28 days after hospital release
  To determine whether, when accompanied by the caregiver, children with severe acute malnutrition (SAM), daily cleaning with wipes containing 2% chlorhexidine gluconate (HCG) reduces the incidence of nosocomial bacteremia suspected and / or confirmed by the laboratory compared to baseline data and compared to daily soap and water cleanup administered by the caregiver.